CLINICAL TRIAL: NCT06429241
Title: A Phase I Clinical Study Evaluating the Distribution and Dynamic Behavior of Nuclide Labeled TH-SC01 Cells in Vivo in Patients With Perianal Fistula
Brief Title: Evaluate the Distribution and Dynamic Behavior of TH-SC01 Cells in Vivo in Patients With Perianal Fistula
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-TH-SC01-I-007
Record Dates: First submitted 2024-05-09; First posted 2024-05-24 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Anal Fistula; Complex Perianal Fistulas; Crohn's Disease
MeSH Terms: conditions — Rectal Fistula; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCs treatment group (Experimental): Intralesional injection of expanded human umbilical cord-derived mesenchymal stem cells suspension.
  Interventions: Biological: Mesenchymal Stem Cells (MSCs)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSCs) — single dose injection (120 million cells)

SUMMARY:
The purpose of this study is to evaluate the distribution and dynamic behavior of Nuclide labeled TH-SC01 cells in vivo in patients with perianal fistula

DETAILED DESCRIPTION:
A Phase I clinical study evaluating the distribution and dynamic behavior of Nuclide labeled TH-SC01 cells in vivo in patients with perianal fistula

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Subjects with Crohn's disease or complex perianal fistula diagnosed at least 6 months earlier according to the Chinese Consensus Opinion on the Diagnosis and Treatment of Inflammatory Bowel Diseases (Beijing, 2018).Subjects with active perianal fistula and non active luminal CD defined by a CDAI ≤ 200.
3. For patients with perianal fistula, 1≤ the number of internal openings ≤2, and 1≤ the number of external openings ≤3, the fistula of the patient needs to be drained smoothly
4. All subjects and their partners were not planning to have a child from screening to the end of the trial and agreed to use effective non-drug contraception during the trial.
5. ECOG score 0~1, ASA grade I~II
6. Subjects failed to respond to adequate treatment with any of the conventional antibiotics, immunomodulatory drugs (including steroids), anti-tumor necrosis factor-α (TNF-α) monoclonal antibodies and other biological agents.

Exclusion Criteria:

1. Subjects with active infection evaluated by the investigator.
2. Subjects with Crohn&#39;s disease requiring immediate therapy.
3. Subjects with abscess or collections &gt;2 cm.
4. Subjects with rectal and/or anal stenosis and/or active proctitis.
5. Subjects who treated with systemic steroids in the 4 weeks prior to stem cells administration.
6. Subjects with abnormal laboratory results: liver function: total bilirubin &gt;=1.5 × ULN, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) &gt;=2 × ULN; renal function: creatinine clearance below 60 mL/minute calculated using Cockcroft-Gault formula or by serum creatinine &gt;=1.5 × upper limit of normal (ULN).
7. Subjects with malignant tumors or a history of malignant tumors.
8. Subjects with severe, progressive, uncontrolled hepatic, hematological, gastrointestinal (except Crohn&#39;s disease), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral diseases.
9. Serum virology test (HBeAg, HCV antibody, HIV antibody, Treponema pallidum antibody) positive.
10. Subjects allergic to Human serum albumin, human platelet lysate, gentamicin sulfate, anesthetic drug
11. Subjects who has received stem cells therapy.
12. Subjects who has major surgery or severe trauma within 6 months prior to the screening period.
13. Subjects who has received any investigational drug within 3 months prior to the screening.
14. Subjects deemed inappropriate by the investigator to participate in this clinical trial.
15. The female participant who is pregnant, or is lactating.
16. Not suitable for PET/CT examination.
17. Participants considered inappropriate to participate in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value | 8-12 hour、32-36 hour、56-60 hour、104-108 hour、152-156 hour，296-300 hour
  Standardized values of organs or tissues after PET/CT imaging after local injection in patients with perianal fistula

SECONDARY OUTCOMES:
Effectiveness endpoint:Proportion of subjects with clinically significant effect at week 24 after local injection | Week 1，Week 4，Week 24
  Change from baseline in pain score (VAS score).Total score ranges from 0 to 10. Higher score means more pain.
Safety endpoint: Treatment-related adverse events/adverse reactions, serious adverse events/serious adverse events | Week 1，Week 4，Week 24，Month 24
  All subjects were observed for any adverse events/reactions or serious adverse events/reactions that occurred during the clinical trial, including but not limited to clinically significant abnormal changes in clinical symptoms, physical examination, vital signs examination, laboratory examination, 12-lead electrocardiogram examination, etc. The clinical features, severity, occurrence time, end time, treatment and outcome of the disease should be recorded, and the correlation between the disease and the investigational drug should be determined.
Radiation exposure: Uptake rate (%ID), absorbed dose, and systemic effective dose in vital organs or tissues after local injection of nuclide labeled TH-SC01 cells. | Week 1
  Based on the image data obtained by PET/CT scan, OLINDA's sphere model was used to delineate the injection site and important organs or tissues as areas of interest (ROI), obtain standardized uptake values (SUV) of each ROI, and obtain time-radioactive activity curves (TACs) of each tissue and organ. The absorbed dose of vital organs or tissues, the equivalent dose of the whole body, and the distribution and change of transplanted cells in different tissues or organs at different time points are described

CONTACTS AND LOCATIONS:
Locations (1):
- The first Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided